CLINICAL TRIAL: NCT01109563
Title: Reaching and Motivating Change in Teen Marijuana Smokers
Brief Title: Teen Marijuana Check-Up
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Denise Walker (Other)
Collaborators: Virginia Polytechnic Institute and State University (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Denise Walker, Principal Investigator, University of Washington
Organization: University of Washington (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 37852-G; 2R01DA014296-09A1 (NIH)
Record Dates: First submitted 2010-04-21; First posted 2010-04-23 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Cannabis Use Disorder
Keywords: cannabis use disorder; marijuana; motivational enhancement treatment; cognitive behavioral treatment; continuing care
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Computer Check-In Control (Active Comparator): The Computer Check-In gives the participant contact with the research therapist, an assessment of marijuana use and the current impact of use, and a reminder about optional support sessions.
  Interventions: Behavioral: Marijuana Check-Ins
- Marijuana Check-Ins (Experimental): The MCI, a MET intervention, will include the provision of personalized feedback with a motivational interviewing style. The focus of these sessions will be individualized to participants based on recent marijuana use and related experiences. Feedback given to participants during the MCI session will review progress toward goals as self-reported in percent days abstinent, normative data regarding marijuana use, review of reported consequences of marijuana use, review of abuse and dependence criteria reported, comparison of consequences and abuse and dependence symptoms reported over time, review of the positive outcomes from reductions in use, and review of immediate and long-term life goals and how their marijuana goal will affect these. HEs will offer particular encouragement to take advantage of CBT sessions to participants who feel they currently need treatment.
  Interventions: Behavioral: Marijuana Check-Ins

INTERVENTIONS:
Behavioral: Marijuana Check-Ins — The MCI, an MET intervention, will include the provision of personalized feedback with a motivational interviewing style. The focus of these sessions will be individualized to participants based on recent marijuana use and related experiences. Feedback given to participants during the MCI session will review progress toward goals as self-reported in percent days abstinent, normative data regarding marijuana use, review of reported consequences of marijuana use, review of abuse and dependence criteria reported, comparison of consequences and abuse and dependence symptoms reported over time, review of the positive outcomes from reductions in use, and review of immediate and long-term life goals and how their marijuana goal will affect these. HEs will offer particular encouragement to take advantage of CBT sessions to participants who feel they currently need treatment.

SUMMARY:
This study will test a behavioral intervention tailored for adolescents who smoke marijuana and have concerns about their use. The study's purpose is to determine whether this intervention (two-sessions of motivational enhancement intervention followed by 12 months of optional skills training) will be more effective in reducing the use of this drug if augmented by three periodic motivational enhancement treatment check-in sessions as compared to three periodic computer-based check-in sessions.

HYPOTHESES: (1) Participants in the motivational enhancement treatment check-ins (MCI) condition will reduce their use of marijuana more than participants in the computer based (Comp) condition and report fewer negative consequences. These differences are expected to be greater at later follow-ups (i.e, 9, 12, and 15 months) after repeated check-ins exert a cumulative effect. (2)Engagement in CBT sessions will be greater for those in the MCI condition and will partially mediate the effect on marijuana related outcome indices. (3) The MCI intervention will lead to increased self-efficacy, and decreased normative perceptions of marijuana use by other teens that will also partially mediate the effect of the intervention.

DETAILED DESCRIPTION:
The goal of this trial is to evaluate the efficacy of an enhanced Teen Marijuana Check-Up protocol to reach and intervene with non-treatment seeking adolescents who use marijuana heavily. Two hundred fifty adolescents who use marijuana heavily will receive a 2-session individual motivational enhancement therapy. All participants will also be offered the opportunity, over a 12-month period, to repeatedly re-initiate marijuana counseling. Participants will be randomly assigned to receive one of two types of periodic follow-up contacts: Motivational interviewing-based Marijuana Check-Ins (MCI) or Computer Based Control (Comp) sessions.

All participants will be reassessed at the 6, 9, 12, and 15-month anniversaries of enrollment. Following their initial motivational enhancement therapy, the 125 experimental condition participants will additionally have a motivational enhancement treatment "check-in" session with their counselor at the 4, 7, and 10-month anniversaries of enrollment intended to reinforce the maintenance of treatment gains and motivate continued success, increase motivation to change for participants who did not meet their marijuana use goals, and/or prompt utilization of cognitive-behavioral treatment (CBT) sessions as needed. The 125 comparison participants will complete a computer based questionnaire at the same time intervals to serve as an attentional control.

ELIGIBILITY:
Inclusion Criteria:

1. age (14-19 years old),
2. grade level (9th through 11th) and
3. marijuana use.

Exclusion Criteria:

Individuals will be excluded if:

1. they are not fluent in English,
2. they have a thought disorder that precludes full participation,
3. they refuse to accept randomization to condition,
4. they are high school seniors.

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 252 (Actual)
Dates: Start 2011-03; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
frequency (number of days) of marijuana use | 60 days
  Global Appraisal of Individual Needs - I (self-report measure)
treatment utilization | 90 days
  Global Appraisal of Individual Needs - I
marijuana abuse/dependence symptoms | 60 days
  Global Appraisal of Individual Needs - I
engagement in cognitive behavioral skills training sessions | 90 days
  Frequency of attendance at optional in-school counseling sessions

SECONDARY OUTCOMES:
self-efficacy | 90 days
  Self-efficacy scale that assesses self-efficacy for avoiding marijuana use
normative perceptions of peer marijuana use | 90 days
  Descriptive perceived norms concerning the frequency of marijuana use by other adolescents of the participant's age

CONTACTS AND LOCATIONS:
Overall Officials: Denise D Walker, PhD, Principal Investigator — University of Washington School of Social Work